CLINICAL TRIAL: NCT03782636
Title: Interleukin-2 Therapy of Autoimmunity in Diabetes (ITAD)
Acronym: ITAD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Clinical Trials Research Unit (OCTRU) (Unknown); Centre for Statistics in Medicine, Oxford (Unknown); Juvenile Diabetes Research Foundation (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13341
Record Dates: First submitted 2018-09-07; First posted 2018-12-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Type1 Diabetes
MeSH Terms: interventions — aldesleukin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aldesleukin (Experimental): Ultra-low dose aldesleukin injected subcutaneously, at a dose of 0.2 x 106 IU/m2 twice-weekly , three days apart, for 6 months.
  Interventions: Drug: Aldesleukin
- Placebo (Placebo Comparator): Placebo sc, at a similar dose (expressed in ml) to the active drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aldesleukin — PROLEUKIN® 18 x 106 IU
  Powder for solution for injection or infusion
  Arms: Aldesleukin
Other: Placebo — sterile diluent used for the aldesleukin preparation and 5% glucose
  Arms: Placebo

SUMMARY:
The main purpose of this study is to see if a drug called aldesleukin, can preserve insulin production in children and young adults recently diagnosed with type 1 diabetes.

One group will receive aldesleukin and the other a placebo.

DETAILED DESCRIPTION:
Investigators know that the longer people with diabetes can produce their own insulin, the better it is for the control of their blood glucose levels and long-term complications.

People get type 1 diabetes because their immune system, the part of the body, which helps fight infections, mistakenly attacks and destroys the beta cells in the pancreas that produce insulin. As the immune system destroys these insulin-producing cells, the body's own ability to produce insulin decreases and diabetes develops.

At diagnosis, there are usually a small number of beta cells (10-20%) left in the pancreas, which still produce small amounts of insulin. This is called 'beta cell function' and it is assessed by measuring C-peptide, which is a protein made by the pancreas when insulin is produced. Most people with type 1 diabetes eventually stop producing insulin themselves, this may occur rapidly in a few months, or more slowly over several years.

New treatments preserving insulin production could improve management of diabetes. This could be done by using drugs acting on cells of the immune system. In type 1 diabetes, there is an imbalance between cells of the immune system, and there is evidence that one protein produced by our body, called Interleukin-2, could help in resetting the balance between those cells. It is important to start this treatment soon after diagnosis because this when there is the best chance of saving the beta cells still left in the pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent to participate or assent with parental consent
2. Be aged 6-18 years
3. Be diagnosed with T1D (Type 1 Diabetes) (at least one autoantibody positive), requiring insulin treatment
4. Be within 6 weeks from diagnosis of T1D (at screening)
5. Have a random C-peptide > 200 pmol/l
6. Normal full blood count

Exclusion Criteria:

1. Non-type 1 diabetes (type 2 or monogenic diabetes) and secondary diabetes
2. Pre-existing autoimmune disease (excluding type 1 diabetes)
3. Hypersensitivity to aldesleukin or any of the excipients
4. History of severe cardiac disease (NYHA Class III or IV)
5. History of malignancy within the past 5 years (with the exception of adequately treated basal or squamous cell carcinoma or cervical carcinoma in situ)
6. Clinically significant abnormal laboratory values (out of range and associated with clinical symptoms or signs) in haematology, biochemistry, thyroid, liver and kidney function
7. Pre-existing severe major organ dysfunction or seizure disorders
8. Participation in another clinical trial (CTIMP) within 4 months prior to screening
9. Females who are pregnant, lactating or intend to get pregnant during the study
10. Females of childbearing potential who are unwilling or unable to comply with contraceptive advice and regular pregnancy testing throughout the trial
11. Sexually active males who are unwilling or unable to comply with contraceptive advice
12. Current use of immunosuppressive agents or steroids
13. Current treatment with hepatotoxic, nephrotoxic, myelotoxic, or cardiotoxic products
14. Active clinical infections - participants can be recruited after a minimum period of 48 h after last day of feeling unwell or last day of antibiotic/anti-viral treatment
15. Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the participant ineligible for inclusion because of a safety concern
16. Children with compliance problems (families where the local investigators consider that problems with compliance may be an issue)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Differences in slopes of DBS (Dried Blood Spot) C-peptide over the 6 month-treatment period between the active and placebo groups. | Weekly DBS C-peptide collected during the 6-month treatment period, and then monthly during the 6 months of follow-up

SECONDARY OUTCOMES:
Change in Treg, Teff and NK56bright cell frequencies and phenotypes from baseline | At baseline and then1, 2 , 3, 6 and 12 months from the beginning of treatment
Safety will be assessed at each visit (reported reactions using CTCAE grading v5.0) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Assessment of the most commonly reported reactions to low- or high-dose aldesleukin, namely influenza-like syndrome, skin reaction, diarrhoea, nausea using CTCAE grading v5.0
Safety will be assessed at each visit (temperature in celsius) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Vital signs - temperature in celsius
Safety will be assessed at each visit (weight, in kilograms) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Vital signs - weight, in kilograms
Safety will be assessed at each visit (blood pressure: systolic/diastolic) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Vital signs - blood pressure: systolic/diastolic
Safety will be assessed at each visit (heart rate: bpm) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Vital signs - heart rate: bpm
Safety will be assessed at each visit (AST, ALT, ALP, GGT units per liter (U/L) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Abnormal laboratory parameters liver function (AST, ALT, ALP, GGT units per liter (U/L)
Safety will be assessed at each visit total bilirubin - milligrams per deciliter (mg/dL) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Abnormal laboratory parameters liver function total bilirubin - milligrams per deciliter (mg/dL)
Safety will be assessed at each visit (urea and creatinine - mmol/L) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Abnormal laboratory parameters kidney function (urea and creatinine - mmol/L)
Safety will be assessed at each visit (full blood count - 109/L) | At screening, baseline and then 1, 2 , 3, 6 and 12 months from the beginning of treatment
  Abnormal laboratory parameters full blood count - 109/L
Changes in the absolute numbers of T, B and NK (Natural Killer) cells. | At baseline and then, 1, 2 , 3, 6 and 12 months from the beginning of treatment
Change in HbA1c and daily insulin requirements during the trial period. | HbA1c - At baseline and then 3,6 and 12 months Insulin dose data -Baseline and then 1, 2, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Johnson, Professor, Principal Investigator — University of Oxford
Locations (5):
- United Kingdom (5):
  - Oxford Children's Hospital, Oxford, Oxfordshire
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - The Great North Children's Hospital, Newcastle upon Tyne
  - Nottingham Children's Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided